CLINICAL TRIAL: NCT00781560
Title: A Cross-sectional Study to Survey the Awareness of Chinese National Adult Lipid Treatment Guideline (2007) and the Rate of Patients (on Treatment) Achieving the Hyperlipidaemia Treatment Goal With Crestor 5mg to 10mg for 8 Weeks
Brief Title: Awareness of Chinese National Adult Lipid Treatment Guideline (2007) and Rate of Patients Achieving the Treatment Goal
Acronym: CRE NIS
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Karen Atkin/ VP. China R&D, AstraZeneca Pharmaceuticals
Other Study IDs: NIS-CCN-CRE-2008/1
Record Dates: First submitted 2008-10-28; First posted 2008-10-29 (Estimated); Last update posted 2009-08-07 (Estimated); Status verified 2009-08

CONDITIONS: Hyperlipidemia
Keywords: Hyperlipidemia; Chinese National Adult Lipid Treatment Guideline (2007); Crestor®
MeSH Terms: conditions — Hyperlipidemias

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: patients being diagnosed as dyslipidemia but not receiving Crestor®
- 2: hypercholesterolemia or mixed dyslipidemia and have been initiated treatment with Crestor®

SUMMARY:
This study is designed to survey the awareness rate of Chinese National Adult Lipid Treatment Guideline (2007) by cardiologists; To survey the control rate of the patients with dyslipidemia in "real world"; and to evaluate the percentage of hyperlipidemia patients who achieved target LDL-C level according to the Chinese National Adult Lipid Treatment Guideline (2007) following 8-week treatment by Crestor® 5mg or 10mg

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as dyslipidemia by doctors
* Having lipids test and record within one months
* Diagnosed as hypercholesterolemia or mixed dyslipidaemias and has been prescribed Crestor® 5mg or 10mg

Exclusion Criteria:

* Unable or unwilling to provide the Inform Consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who has been diagnosed as hypercholesterolemia and decided by physician to use Crestor® 5mg or 10mg or other regimens (TLC or other lipid-lowering agents)
Sampling Method: Non-Probability Sample
Enrollment: 2575 (Actual)
Dates: Start 2008-10; Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
the awareness rate of Chinese National Adult Lipid Treatment Guideline (2007) by cardiologists | 1 time
the control rate of patients reaching target LDL-C level | 8 weeks

SECONDARY OUTCOMES:
the percent change from baselines in TC, TG, HDL-C | 8 weeks
the percentage of hyperlipidemia patients in different risk categories who achieved target LDL-C level according to the Chinese National Adult Lipid Treatment Guideline (2007) | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Karen Atkin, Study Director — Astrazeneca China R&D; Zhu Junren, Principal Investigator — Fudan University
Locations (15):
- China (15):
  - Research Site, Beijing, Beijing Municipality
  - Research Site, Chenzhen, Guangdong
  - Research Site, Guangzhou, Guangdong
  - Research Site, Harbin, Heilongjiang
  - Research Site, Zhengzhou, Henan
  - Research Site, Nanjing, Jiangsu
  - Research Site, Shenyang, Liaoning
  - Research Site, Jinan, Shandong
  - Research Site, Qingdao, Shandong
  - Research Site, Shanghai, Shanghai Municipality
  - Research Site, Xi’an, Shanxi
  - Research Site, Chengdu, Sichuan
  - Research Site, Tianjin, Tianjin Municipality
  - Research Site, Hangzhou, Zhejiang
  - Reseearch Site, Ningbo, Zhejiang